CLINICAL TRIAL: NCT02884492
Title: Imaging Tau in Alzheimer's Disease and Normal Aging
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped due to published data regarding THK-5351 non-specificity in Tau imaging
Sponsor: William Charles Kreisl (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, William Charles Kreisl, Principal Investigator, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAQ7868; 1K23AG052633-01 (NIH)
Record Dates: First submitted 2016-08-25; First posted 2016-08-31 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer's Disease
Keywords: inflammation; aging; mild cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Inflammation; Cognitive Dysfunction | interventions — THK5351; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cognitive impairment (Experimental): Adults with Alzheimer's disease, preclinical Alzheimer's disease or impairment due to suspected non-Alzheimer's disease pathophysiology will receive 18F-THK- 5351 and/or lumbar puncture (optional).
  Interventions: Drug: 18F-THK-5351; Procedure: Lumbar Puncture (optional)
- No cognitive impairment (Active Comparator): Normal aging adults will receive 18F-THK- 5351 and/or lumbar puncture (optional).
  Interventions: Drug: 18F-THK-5351; Procedure: Lumbar Puncture (optional)

INTERVENTIONS:
Drug: 18F-THK-5351 — 18F-THK-5351 is a PET radioligand that binds abnormal tangles made of the protein tau. These tau tangles develop in the brain in people with Alzheimer's disease.
  Other Names: [18F] THK5351
Procedure: Lumbar Puncture (optional) — Subjects have the option to have lumbar puncture performed for the measurement of Alzheimer's disease biomarkers in cerebrospinal fluid.

SUMMARY:
This study is being done to learn about tau tangles in Alzheimer's disease. A type of PET scan is used to measure the abnormal accumulation of protein called tau in the brain. These are thought to be involved in Alzheimer's disease. The investigators will also perform brain MRI and to tests to measure the participant's memory and thinking.

DETAILED DESCRIPTION:
This study is being done to determine the relationship between tau tangles and cognitive impairment in elderly subjects with different clinical and biomarker profiles of Alzheimer's disease (AD). Subjects will undergo screen that includes neuropsychological testing and brain MRI. This study uses a special type of scan called a PET scan to take pictures of the brain. During the PET scan, a special radioactive dye called 18F-THK-5351 is injected into the body. 18F-THK-5351 sticks to abnormal tangles made of the protein tau. Subjects will have the option to have lumbar puncture performed to measure CSF concentrations of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older.
2. Meet criteria for either a) amnestic mild cognitive impairment (single or mixed domain) or mild Alzheimer's disease, or b) have no cognitive impairment, based on history, exam, neuropsychological testing, and consensus diagnosis. MCI and mild AD patients must have Clinical Dementia Rating scale score of 0.5 or 1. Unimpaired subjects must have Clinical Dementia Rating scale score of 0.
3. Subjects unable to provide informed consent must have a surrogate decision maker.
4. Written and oral fluency in English or Spanish.
5. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
6. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain brain disorders other than MCI or AD.
2. Certain significant medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Contraindication to MRI scanning.
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. History of kidney disease or presence of impaired kidney function based on laboratory tests at the screening visit.
6. History of liver disease or presence of impaired liver function based on laboratory tests at the screening visit.
7. Participation in the last year in a clinical trial for a disease-modifying drug for AD.
8. Inability to have a catheter in subject's vein for the injection of radioligand.
9. Inability to have blood drawn from subject's veins.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Kreisl, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Impairment | No Cognitive Impairment
Started | 7 | 10
Completed | 7 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Impairment | No Cognitive Impairment | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 6 | 7 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: 18F-THK-5351 Standardized Uptake Value Ratio
Description: The standardize uptake value ratio is the concentration of radioactivity measured from the 18F-THK-5351 PET scan in the posterior cingulate gyrus, divided by that in the cerebellar gray matter (the reference region, which is expected to be devoid of tau pathology). This ratio is a relative measure of 18F-THK-5351 binding, and therefore of tau pathology, in brain tissue. PET image data was acquired from 50 min post-injection to 70 min post-injection of 18F-THK-5351.
Time Frame: PET image data collected 50 min post-injection to 70 min post-injection of 18F-THK-5351
Measure: Median (Full Range); unit: Standardized uptake value ratio
Arm/Group | Cognitive Impairment | No Cognitive Impairment
Number analyzed (Participants) | 7 | 10
Standardized uptake value ratio | 1.78 [1.41 to 2.04] | 1.44 [1.08 to 1.56]

ADVERSE EVENTS:
Time Frame: Up to 24 hours after the PET scan for follow up adverse event reporting
Arm/Group | Cognitive Impairment | No Cognitive Impairment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. THK-5351 has been found to bind to monoamine oxidase B as well as to tau aggregates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02884492/Prot_SAP_000.pdf